CLINICAL TRIAL: NCT02350244
Title: Active Prevention of MSDs (Musculoskeletal Disorders, Upper and Spine Members) in the Context of Computer Screen Work
Acronym: I-Preventive
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None
Other Study IDs: CHU-0219
Record Dates: First submitted 2015-01-13; First posted 2015-01-29 (Estimated); Last update posted 2015-01-29 (Estimated); Status verified 2015-01

CONDITIONS: Symptomatic Musculoskeletal Diseases; Latent Musculoskeletal Diseases
Keywords: musculoskeletal diseases; eyestrain; occupational diseases; computer work; muscle stretching exercise; computer software application; MSDs
MeSH Terms: conditions — Musculoskeletal Diseases; Asthenopia; Occupational Diseases

ARMS (2):
- Experimental group (Experimental): Subjects of the experimental group will have to follow an intervention for one month, consisting in active breaks from computer work
  Interventions: Behavioral: Computer program
- Control group (Other): Control group patients had no intervention
  Interventions: Behavioral: Computer program

INTERVENTIONS:
Behavioral: Computer program — Intervention consists in a computer program suggesting workers to take active breaks at given times of their working day, during one month.

SUMMARY:
Evaluate the benefit of an intervention by a computer program comprising active breaks, in the form of a personalized self-program on functional impairment and / or pain, among employees with latent or symptomatic upper extremity MSDs and spine (+/- eyestrain) in connection with the computer work environment.

DETAILED DESCRIPTION:
The benefit of the intervention will be assessed among four groups of subjects: symptomatic and asymptomatic subjects randomized in control or experimental group.

Subjects of the experimental group will have to follow an intervention for one month, consisting in active breaks from computer work. Control group patients had no intervention.

Symptoms of MSD will be assessed via questionnaire before and after intervention, in all groups.

ELIGIBILITY:
Inclusion Criteria:

* - To carry out a professional activity.
* To be involved in a computer work for at least 5 hours a day.
* To be between 18 and 65 years.

Exclusion Criteria:

* - To be in sick leave.
* Rheumatic and neurological diseases which needed treatment.
* Workstations which have been recently changed.
* A behavioral and/or comprehension trouble

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2014-06; Primary Completion 2014-11 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Nordic style questionnaire score | at 1 month

SECONDARY OUTCOMES:
Evolution of " Nordic style " and eyestrain questionnaires | at 1 month
Evolution of global psychological status (HAD) | at 1 month
Evolution of psychosocial work characteristics (VAS stress and satisfaction at work) | at 1 month
Occurrence sick leave and frequency of work trips during the study. | at 1 month
Adherence to the self-program | at 1 month

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de Clermont-Ferrand, Clermont-Ferrand, France

REFERENCES:
- [Derived] Lanhers C, Pereira B, Garde G, Maublant C, Dutheil F, Coudeyre E. Evaluation of 'I-Preventive': a digital preventive tool for musculoskeletal disorders in computer workers-a pilot cluster randomised trial. BMJ Open. 2016 Sep 22;6(9):e011304. doi: 10.1136/bmjopen-2016-011304. PMID 27660316